CLINICAL TRIAL: NCT07207980
Title: Lifestyle Intervention Clinical Trial for the Remission of Type 2 Diabetes Mellitus in Primary Care (CREDOenAP)
Brief Title: Lifestyle Intervention for Type 2 Diabetes in Primary Care (CREDOenAP)
Acronym: CREDOenAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc Sanitari Pere Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREDOenAP
Record Dates: First submitted 2025-09-16; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 Diabetes Mellitus (T2DM); Diabetes Remission; Lifestyle Intervention; Primary Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The program consists of biweekly in-person and telephone visits, focused on implementing a personalized dietary plan with carbohydrate restriction, based on the American Diabetes Association recommendations; moderate and accessible physical activity; circadian rhythm regularization; and psychological counseling and support.
  Interventions: Behavioral: CREDOenAP intervention
- Control group (No Intervention): They will receive the standard clinical treatment for diabetes

INTERVENTIONS:
Behavioral: CREDOenAP intervention — Intervention program with intensive lifestyle counseling, added to standard pharmacological treatment subsequently adjusted according to clinical needs and outcomes. The intervention will last 6 months and consists of biweekly in-person and telephone visits. Patients will follow a personalized dietary plan with carbohydrate restriction, based on the recommendations of the American Diabetes Association; engage in moderate and accessible physical activity; implement circadian rhythm regularization; and receive psychological counseling and support.
  Arms: Intervention group

SUMMARY:
The purpose of this clinical trial is to determine whether an intensive lifestyle intervention can achieve remission of type 2 diabetes mellitus (T2DM) in adult patients treated in primary care. The main questions the study seeks to answer are:

* What proportion of participants achieve diabetes remission after 6 months of intervention?
* How many participants maintain remission 12 months after completing the program (18 months total)?

Participants will:

* Follow a personalized dietary plan with carbohydrate restriction.
* Engage in moderate, accessible physical activity.
* Implement strategies to improve circadian rhythm regularity.
* Receive psychological counseling and support.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Men and women aged 18-80 years, inclusive.
3. Confirmed diagnosis of T2DM according to recognized diagnostic criteria
4. Most recent recorded hemoglobin A1c (HbA1c) > 6.5%.
5. Body Mass Index (BMI) greater than 27 kg/m².

Exclusion Criteria:

1. Failure to meet the diagnostic criteria for T2DM in the screening laboratory tests.
2. Being dependent for basic activities of daily living (Barthel score ≤ 90 points).
3. Lack of willingness to cooperate with the follow-up of the lifestyle intervention plan.
4. Presence of serious or terminal comorbidities significantly worsening short- to medium-term prognosis (active cancer, terminal chronic diseases, myocardial infarction within the last 6 months, acute heart failure or NYHA stage ≥ III, etc.).
5. History of ketoacidosis.
6. Presence of criteria or potential autoimmune insulinopenia (abnormal C-peptide, anti-GAD+ antibodies, pattern of basal and/or glucose-stimulated hypoinsulinemia).
7. Cognitive impairment.
8. Weight loss exceeding 5 kg in the past 6 months.
9. Significant changes in physical activity and/or dietary patterns in the past 6 months.
10. History of eating disorders.
11. History of substance abuse.
12. History of severe psychiatric disorders.
13. Pregnancy or intention to become pregnant within the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-11 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-11 (Estimated)

PRIMARY OUTCOMES:
Presence of T2DM remission | After 6 months of intervention and 12 months after the intervention
  Glycated hemoglobin (HbA1c): T2DM remission will be considered if HbA1c is < 6.5% after 6 months of intervention and at least 3 months without antidiabetic medication. HbA1c will be determined by blood analysis after a minimum of 8 hours of fasting
  Fasting plasma glucose: T2DM remission will be considered if fasting venous plasma glucose is < 126 mg/dL after 6 months of intervention and at least 3 months without antidiabetic medication. Fasting plasma glucose will be measured by venous blood analysis after a minimum of 8 hours of fasting

SECONDARY OUTCOMES:
Blood pressure | After 6 months of intervention and 12 months after the intervention.
  Blood pressure will be measured three times after the participant has been seated at rest for 10 minutes with uncrossed legs. The mean of the last two measurements will be used for statistical analysis. Systolic and diastolic blood pressure will be reported in mmHg using a brachial cuff sphygmomanometer.
Total cholesterol | After 6 months of intervention and 12 months after the intervention
  Measured in mg/dL via blood analysis.
HDL cholesterol | After 6 months of intervention and 12 months after the intervention
  High-density lipoprotein (HDL) cholesterol measured in mg/dL via blood analysis.
LDL cholesterol | After 6 months of intervention and 12 months after the intervention
  Low-density lipoprotein (LDL) cholesterol measured in mg/dL via blood analysis.
Apolipoprotein B100 (ApoB100) | After 6 months of intervention and 12 months after the intervention
  A protein involved in cholesterol transport and relevant for evaluating elevated cholesterol causes, measured in mg/dL via blood analysis.
Triglycerides | After 6 months of intervention and 12 months after the intervention
  Measured in mg/dL via blood analysis
Presence and size of atherosclerotic plaques in carotid arteries | After 6 months of intervention and 12 months after the intervention
  Assessed via Doppler ultrasound of the supraaortic trunks. If plaques are present, the total plaque area will be measured in cm², and changes in plaque area will be tracked throughout the study.
Weight | After 6 months of intervention and 12 months after the intervention
  Measured in kilograms (kg)
Body Mass Index (BMI) | After 6 months of intervention and 12 months after the intervention
  Calculated from weight and height using the formula: BMI = weight (kg) / [height (m)]².
Abdominal circumference | After 6 months of intervention and 12 months after the intervention
  Measured at the midpoint between the lowest rib and the iliac crest during maximal inspiration and expiration, in centimeters (cm)
Insulin resistance | After 6 months of intervention and 12 months after the intervention
  Evaluated using the HOMA-IR index (Homeostasis Model Assessment of Insulin Resistance), which estimates insulin resistance and beta-cell function. Determined via blood analysis after a minimum 8-hour fast. Values above 2.5 may indicate T2D. Calculated as: [fasting insulin (μU/mL) x glucemia basal (mmol/L)] / 22.5 = [fasting insulin (μU/mL) x (Glucemia basal (mg/dL) x 0,0555)] / 22.5
Pancreatic activity | After 6 months of intervention and 12 months after the intervention
  Assessed using the HOMA-B index, which evaluates the function and activity of pancreatic beta cells. HOMA-B, together with HOMA-IR, helps in the diagnosis of T2D. Values between 167 and 175 are considered normal and not indicative of T2D. Values below this range suggest impaired beta-cell function, resulting in insufficient insulin production (insulinopenia).
Fasting insulin | After 6 months of intervention and 12 months after the intervention
  Measures the amount of insulin in a blood sample. Insulin is a hormone produced by the pancreas. Normal values range between 5-25 U/mL. It will be measured via blood analysis after a minimum 8-hour fast.
Metabolic Syndrome Diagnosis | After 6 months of intervention and 12 months after the intervention
  Metabolic Syndrome Diagnosis is established if at least three of the following five criteria are present:
  * Abdominal circumference: Men of European descent > 94 cm; Women of European descent > 80 cm. For other ethnicities, cut-off points are defined according to the International Diabetes Federation (IDF). (López De La Torre et al., 2010)
  * Fasting glucose: > 100 mg/dL or receiving pharmacological treatment for hyperglycemia.
  * Triglycerides: > 150 mg/dL or receiving lipid-lowering therapy.
  * HDL cholesterol: < 40 mg/dL in men; < 50 mg/dL in women, or receiving lipid-lowering therapy.
  * Blood pressure: Systolic > 130 mmHg or Diastolic > 85 mmHg, or receiving antihypertensive treatment.
NAFLD Liver Fat Score | After 6 months of intervention and 12 months after the intervention
  Non-alcoholic fatty liver disease (NAFLD) is a condition characterized by excessive fat accumulation in the liver. Its severity can vary according to the score: < -1.455 low risk, -1.455 to 0.675 intermediate risk, > 0.675 high risk (Angulo et al., 2007; Kotronen et al., 2009).
  The calculation is determined using the following formula:
  -2.89 + 1.18 × Metabolic Syndrome (Yes = 1 / No = 0) + 0.45 × T2DM (Yes = 2 / No = 0) + 0.15 × Fasting Insulin (mU/L) + 0.04 × Fasting Serum AST (U/L) - 0.94 × AST/ALT ratio
NAFLD Fibrosis Score | After 6 months of intervention and 12 months after the intervention
  The identification and quantification of fibrosis are clinically relevant since fibrosis is associated with an unfavorable clinical prognosis. An NFS > 0.676 indicates the presence of advanced fibrosis (Angulo et al., 2007; Kotronen et al., 2009). The calculation is determined using the following formula:
  -1.675 + 0.037 × Age (years) + 0.094 × BMI (kg/m²) + 1.13 × IFG/diabetes (Yes = 1 / No = 0) + 0.99 × AST/ALT ratio - 0.013 × Platelets (×10⁹/L) - 0.66 × Albumin (g/dL)
Physical activity | After 6 months of intervention and 12 months after the intervention
  Physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ)
Nutritional and energy composition: | After 6 months of intervention and 12 months after the intervention
  The 24-hour dietary recall questionnaire will be administered at each biweekly visit
Smoking habits | After 6 months of intervention and 12 months after the intervention
  Measured by a study-specific questionnaire
Alcohol consumption | After 6 months of intervention and 12 months after the intervention
  Alcohol intake will be quantified using a questionnaire combined with a standardized alcohol unit conversion calculator
Circadian habits | After 6 months of intervention and 12 months after the intervention
  Measured by a study-specific questionnaire
Health status | After 6 months of intervention and 12 months after the intervention
  SF-36: This is a generic scale that provides a health status profile and is applicable both to patients and to the general population
Medication consumption | After 6 months of intervention and 12 months after the intervention
  Defined Daily Dose (DDD) by active substance: DDDs of the active substances consumed will be classified according to ATC7. Each ATC classification has a defined daily dose based on international standards, which determine the recommended maximum daily amount for the approved indication of the active substance
Number of hypoglycemia episodes | During each follow-up telephone visit throughout the intervention, after 6 months of intervention and 12 months after the intervention
  Episodes of hypoglycemia detected by patients through capillary blood glucose levels and/or recorded in eCAP during the intervention (plasma glucose <60 mg/dl)
Number of symptomatic hyperglycemia episodes | During each follow-up telephone visit throughout the intervention, after 6 months of intervention and 12 months after the intervention
  Episodes of hyperglycemia recorded in eCAP during the intervention (plasma glucose >350 mg/dl accompanied by compatible symptoms such as general malaise, nausea, asthenia, among others)
Total number of healthcare visits | During each follow-up telephone visit throughout the intervention, after 6 months of intervention and 12 months after the intervention
  Annual contacts with the healthcare system including Primary Care (physicians and nursing), Specialized Care, and Emergency Care
Number of diabetes-related emergency episodes | During each follow-up telephone visit throughout the intervention, after 6 months of intervention and 12 months after the intervention
  Emergency visits related to diabetes during the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Ternianov, Principal Investigator — Parc Sanitari Pere Virgili
Locations (1):
- Parc Sanitari Pere Virgili, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-09-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT07207980/Prot_000.pdf